CLINICAL TRIAL: NCT00584961
Title: BIMET Study: Evolution of Metabolic and Cardiovascular Risks Factors in Patients With Bipolar Disorder
Acronym: BIMET
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1281161
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Bipolar Disorder
Keywords: Metabolic Syndrome, Bipolar Disorder and Cardiovascular Risk Factors
MeSH Terms: conditions — Bipolar Disorder; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 600 patients: Patients with diagnosis of Bipolar Disorder (DSM-IV TR)
  Interventions: Other: non-interventional

INTERVENTIONS:
Other: non-interventional — non-interventional

SUMMARY:
To assess the prevalence of Metabolic Syndrome in Spanish population with Bipolar I or II Disorder.

To analyse the clinical progress disease in patients with Bipolar I or II Disorder for 12 months using the assessment of the symptoms disease and the progress of metabolic and cardiovascular risk.

To analyse the health status, quality of life and functioning/disability of patients.

DETAILED DESCRIPTION:
Consecutive patient sampling. In any investigational site, five consecutive patients with diagnosis of Bipolar Disorder will be enrolled in the study

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of Bipolar Disorder (DSM-IV TR)
* Patients or their legal representatives have provided informed consent

Exclusion Criteria:

* Patients are unable to complete or to understand health questionnaires in Spanish language
* Patients enrolled in clinical trials or other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample. Patients >17 years older with diagnosis of Bipolar Disorder (DSM-IV TR)
Sampling Method: Probability Sample
Enrollment: 553 (Actual)
Dates: Start 2007-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Evolution of Modifiable Metabolic and Cardiovascular Risk Factors (Weight, and serum levels of Glucose, Total Cholesterol, LDL-Cholesterol, HDL-Cholesterol and Triglycerides) | 12 months
Clinical Evolution of the Disease | 12 months
Cardiovascular Risk | 12 months

SECONDARY OUTCOMES:
Current pattern of treatment in Bipolar Disorder | 12 month
Prevalence of Metabolic Syndrome in Spanish Population with Bipolar Disorder | 1 day
Patient functional impairment | 12 months
Patient quality of life | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281161&StudyName=BIMET%20Study%3A%20Evolution%20of%20Metabolic%20and%20Cardiovascular%20Risks%20Factors%20in%20Patients%20with%20Bipolar%20Disorder%20